CLINICAL TRIAL: NCT06727604
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2b Study to Assess the Efficacy, Safety, and Tolerability of IMVT-1402 as Treatment for Adult Patients With Graves' Disease
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of IMVT-1402 as Treatment for Adult Participants With Graves' Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMVT-1402-2502; 2024-516020-33-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-09; First posted 2024-12-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Graves' Disease
Keywords: IMVT-1402; Anti Thyroid Drug; Hyperthyroidism; Autoimmune thyroid disease
MeSH Terms: conditions — Graves Disease; Hyperthyroidism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 Period 1 and 2: IMVT-1402 (Experimental)
  Interventions: Drug: IMVT-1402
- Group 2 Period 1 and 2: IMVT-1402 (Experimental)
  Interventions: Drug: IMVT-1402
- Group 2 Period 1: IMVT-1402 and Period 2: Placebo (Experimental)
  Interventions: Drug: IMVT-1402
- Group 3 Period 1 and 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMVT-1402 — 600 mg SC QW for 52 weeks
  Arms: Group 1 Period 1 and 2: IMVT-1402; Group 2 Period 1 and 2: IMVT-1402
Drug: IMVT-1402 — 600 mg SC QW for 26 weeks followed by Placebo SC QW for 26 weeks
  Arms: Group 2 Period 1: IMVT-1402 and Period 2: Placebo
Drug: Placebo — SC QW for 52 weeks
  Arms: Group 3 Period 1 and 2: Placebo

SUMMARY:
This is a study to assess the efficacy, safety, and tolerability of IMVT-1402 in adult participants with Graves' disease (GD) who are hyperthyroid despite antithyroid drug (ATD) treatment.

The primary objective of this study is to evaluate the efficacy of IMVT-1402 versus placebo as assessed by T3 (total triiodothyronine [T3] or free triiodothyronine [FT3]), free thyroxine (FT4), thyroid-stimulating hormone (TSH), and ATD dose at Week 26.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the ability to understand the requirements of the trial, provide written informed consent, and comply with the trial protocol procedures.
* Male or female participants aged ≥ 18 years.
* Participants with diagnosis of GD who are hyperthyroid despite ATD treatment.
* Other, more specific inclusion criteria are defined in the protocol.

Exclusion Criteria:

* Have previously been successfully treated with radioactive iodine (RAI) therapy or have undergone total thyroidectomy.
* Have an autoimmune disease other than GD requiring treatment that, in the Investigator's judgment, puts the participant at undue risk.
* Have moderate-to-severe active thyroid eye disease (TED) and are expected to require immediate surgical intervention and/or are planning corrective surgery/irradiation or medical therapy for TED during study participation.
* Additional exclusion criteria are defined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who are euthyroid (local laboratory T3 [Total T3 or FT3], FT4, and TSH values within normal limits) and off ATD at Week 26 | Week 26

SECONDARY OUTCOMES:
Percentage of participants who are euthyroid and off ATD at Week 52 | Week 52
Percentage of participants who are euthyroid, off ATD, and seronegative for TRAb at Week 52 | Week 52
Percentage of participants who are euthyroid and off ATD at Week 52 and remain euthyroid, off IMVT-1402, and off ATD for 6 months from Week 52 to Week 78 | Week 78
Percentage of participants who are euthyroid and off ATD at Week 52 and remain euthyroid, off IMVT-1402, and off ATD for 12 months from Week 52 to Week 104 | Week 104
Percentage of participants who have a TRAb value a specified amount and are euthyroid and off ATD at Week 26 and remain euthyroid, off IMVT-1402, and off ATD for 6 months from Week 26 to Week 52 | Week 52
Percentage of participants who have a TRAb value a specific amount and are euthyroid and off ATD at Week 26 and remain euthyroid, off IMVT-1402, and off ATD for 12 months from Week 26 to Week 78 | Week 78
Percentage of participants who have T3 (Total T3 or FT3) and FT4 < ULN at Week 2 in participants who have T3 (Total T3 or FT3) and/or FT4 > ULN at baseline | Week 2
Percentage of participants who have T3 (Total T3 or FT3) and FT4 < ULN at Week 4 in participants who have T3 (Total T3 or FT3) and/or FT4 > ULN at baseline | Week 4
Percentage of participants who are euthyroid, off ATD, and seronegative for TRAb at Week 26 | Week 26
Percentage of participants who have T3 (Total T3 or FT3) and FT4 < ULN and are off ATD at Week 26 | Week 26
Percentage of participants who have T3 (Total T3 or FT3) and FT4 < ULN and are off ATD at Week 52 | Week 52

CONTACTS AND LOCATIONS:
Locations (112):
- United States (46):
  - Site Number - 1032, Phoenix, Arizona
  - Site Number - 1036, Phoenix, Arizona
  - Site Number - 1001, Los Angeles, California
  - Site Number - 1062, Orange, California
  - Site Number - 1034, San Francisco, California
  - Site Number - 1035, Santa Clarita, California
  - Site Number - 1005, Torrance, California
  - Site Number - 1006, Walnut Creek, California
  - Site Number - 1013, Englewood, Colorado
  - Site Number - 1010, Newark, Delaware
  - Site Number - 1040, Washington D.C., District of Columbia
  - Site Number - 1029, Clearwater, Florida
  - Site Number - 1055, Jacksonville, Florida
  - Site Number - 1056, Jacksonville, Florida
  - Site Number - 1028, Miami, Florida
  - Site Number - 1011, Orlando, Florida
  - Site Number - 1016, Port Charlotte, Florida
  - Site Number - 1012, West Palm Beach, Florida
  - Site Number - 1038, Atlanta, Georgia
  - Site Number - 1053, Macon, Georgia
  - Site Number - 1020, Stockbridge, Georgia
  - Site Number - 1027, Indianapolis, Indiana
  - Site Number - 1045, Bowling Green, Kentucky
  - Site Number - 1022, New Orleans, Louisiana
  - Site Number - 1048, Shreveport, Louisiana
  - Site Number - 1023, Baltimore, Maryland
  - Site Number - 1026, Boston, Massachusetts
  - Site Number - 1018, Farmington Hills, Michigan
  - Site Number - 1008, Rochester, Minnesota
  - Site Number - 1017, Omaha, Nebraska
  - Site Number - 1007, Las Vegas, Nevada
  - Site Number - 1051, Asheville, North Carolina
  - Site Number - 1057, Canton, Ohio
  - Site Number - 1003, Portland, Oregon
  - Site Number - 1033, Philadelphia, Pennsylvania
  - Site Number - 1015, Summerville, South Carolina
  - Site Number - 1042, Chattanooga, Tennessee
  - Site Number - 1002, Austin, Texas
  - Site Number - 1019, Dallas, Texas
  - Site Number - 1031, Dallas, Texas
  - Site Number - 1025, Houston, Texas
  - Site Number - 1004, Mesquite, Texas
  - Site Number - 1009, Round Rock, Texas
  - Site Number - 1014, San Antonio, Texas
  - Site Number - 1052, San Antonio, Texas
  - Site Number - 1030, Salt Lake City, Utah
- Belgium (3):
  - Site Number - 5303, Antwerp
  - Site Number - 5301, Bruges
  - Site Number - 5302, Brussels
- Georgia (11):
  - Site Number - 8002, Batumi
  - Site Number - 8007, Batumi
  - Site Number - 8006, Kutaisi
  - Site Number - 8008, Marneuli
  - Site Number - 8009, Tbilisi
  - Site Number - 8004, Tbilisi
  - Site Number - 8005, Tbilisi
  - Site Number - 8001, Tbilisi
  - Site Number - 8003, Tbilisi
  - Site Number - 8011, Tbilisi
  - Site Number - 8010, Tbilisi
- Germany (3):
  - Site Number - 6505, Dresden, Saxony
  - Site Number - 6508, Munich
  - Site Number - 6502, Schwerin
- Hungary (6):
  - Site Number - 7558, Békéscsaba
  - Site Number - 7554, Budapest
  - Site Number - 7556, Budapest
  - Site Number - 7557, Debrecen
  - Site Number - 7551, Pécs
  - Site Number - 7552, Szeged
- Italy (12):
  - Site Number - 6004, Bologna
  - Site Number - 6012, Cagliari
  - Site Number - 6011, Genova
  - Site Number - 6002, Milan
  - Site Number - 6009, Milan
  - Site Number - 6007, Milan
  - Site Number - 6010, Napoli
  - Site Number - 6003, Pisa
  - Site Number - 6001, Pisa
  - Site Number - 6005, Roma
  - Site Number - 6013, Siena
  - Site Number - 6008, Varese
- Poland (7):
  - Site Number - 3006, Gliwice
  - Site Number - 3002, Krakow
  - Site Number -3003, Krakow
  - Site Number - 3005, Lublin
  - Site Number - 3004, Lublin
  - Site Number - 3007, Poznan
  - Site Number - 3001, Warsaw
- Puerto Rico (2):
  - Site Number - 1058, San Juan
  - Site Number - 1037, San Juan
- Spain (9):
  - Site Number - 7104, Badalona, Barcelona
  - Site Number - 7109, Barcelona
  - Site Number - 7103, Barcelona
  - Site Number - 7102, Córdoba
  - Site Number - 7106, Granada
  - Site Number - 7105, Madrid
  - Site Number - 7107, Pamplona
  - Site Number - 7108, Pamplona
  - Site Number - 7101, Seville
- United Kingdom (13):
  - Site Number - 7013, Birmingham, England
  - Site Number - 7012, Bristol, England
  - Site Number - 7011, Coventry, England
  - Site Number - 7007, London, England
  - Site Number - 7002, Cardiff
  - Site Number - 7008, Edinburgh
  - Site Number - 7005, Huddersfield
  - Site Number - 7004, Hull
  - Site Number - 7003, London
  - Site Number - 7006, Manchester
  - Site Number - 7001, Newcastle upon Tyne
  - Site Number - 7009, Norwich
  - Site Number - 7010, Nuneaton

IPD SHARING:
Plan to Share IPD: No